CLINICAL TRIAL: NCT07342920
Title: Study of the Prevalence of Active/Passive Smoking and Vaping Among Patients With Cystic Fibrosis
Acronym: Taba-Muco
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9813
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Smoking, Vaping
MeSH Terms: conditions — Cystic Fibrosis; Smoking; Vaping

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the collective unconscious, a patient with cystic fibrosis does not smoke. This belief is so deeply rooted that there is virtually no French data on the prevalence of smoking among this vulnerable population.

Faced with a cohort of patients undergoing a complete transformation (improved quality of life and life expectancy, fewer hospitalizations, reduced respiratory symptoms, better social integration), it is becoming urgent to assess the current situation in order to optimize tobacco prevention.

This is all the more important given the emergence of international studies objectively examining the interactions between smoking, vaping, and the efficacy of Kaftrio.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* With confirmed cystic fibrosis
* Regular follow-up at the Strasbourg Adult Cystic Fibrosis Center

Exclusion Criteria:

* Patients who have undergone a double lung transplant for cystic fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with confirmed cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of smoking in adults with cystic fibrosis | Up to 12 months
  The proportion of adults with cystic fibrosis who smoke:
  Example:
  If 10 out of 100 adults with cystic fibrosis smoke, then the prevalence of smoking in this group is 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - CHU de Strasbourg - France, Strasbourg, France